CLINICAL TRIAL: NCT00330889
Title: A Study of the Pharmacodynamic Effects of Prednisolone on Whole Blood Protein and Gene Expression in Rheumatoid Arthritis Patients
Brief Title: Effects Of Prednisolone On Rheumatoid Arthritis Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 999920/040
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will assess the Pharmacokinetic (PK) and Pharmacodynamic (PD) effects of Prednisolone on Rheumatoid Arthritis (RA) patients.

ELIGIBILITY:
Inclusion criteria:

* Meet the ACR criteria for diagnosis of rheumatoid arthritis.
* Required treatment with Prednisolone.
* Currently on a non-steroidal anti-inflammatory agent (NSAID).
* Willing to stay on current dose of NSAID for two weeks during study.

Exclusion criteria:

* Major health issues such as osteoporosis, diabetes, heart failure, heart attack, kidney failure, or acute infection.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A Study of the Pharmacodynamic Effects of Prednisolone on Whole Blood Protein and Gene Expression in Rheumatoid Arthritis Patients and pharmacodynamic effects on whole blood gene and protein expression.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Modified Disease Activity Score (DAS28), which was composed of swollen and tender joint counts at 28 sites, a patient's global assessment of disease activity using a visual analogue scale (VAS), and ESR. | 14 days
The levels of selected markers of inflammation, which could include (but were not limited to) ESR, C-reactive protein (CRP), interleukin-6 (IL-6), Rheumatoid factor (RF), and soluble tumor necrosis factor-receptor (TNF-R) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (4):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Philadelphia, Pennsylvania
- GSK Investigational Site, Winnipeg, Manitoba, Canada
- GSK Investigational Site, Sheffield, United Kingdom